CLINICAL TRIAL: NCT05806749
Title: Use of the Immunomodulating Agent Belumosudil (KD025) After Combined Kidney and Hematopoeitic Stem Cell Transplantation to Induce Transplant Tolerance: A Pilot Study
Brief Title: Immunological Tolerance in Patients With Mismatched Kidney Transplants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Erik Lum, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mismatch-Tolerance
Record Dates: First submitted 2023-02-01; First posted 2023-04-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: End Stage Kidney Disease; Immunological Tolerance; Kidney Transplant Failure and Rejection; Chronic Kidney Diseases
Keywords: Immunological Tolerance; Kidney Transplant; Tolerance; End Stage Kidney Disease; End Stage Renal Disease; Chronic Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Rejection, Psychology; Renal Insufficiency, Chronic | interventions — CD3 Complex; belumosudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immune tolerance in mismatched kidney transplant recipient (Experimental): Our goal is to establish this regimen as a novel, safe and effective approach for induction of transplant tolerance in HLA single haplotype-matched related and HLA mismatched unrelated recipients of combined Hematopoietic Stem Cell Transplant(HSCT)/ Kidney Transplant (KT). Patients will undergo conditioning with rATG and TLI, followed by infusion of hematopoeitic stem cells from the same donor, a triple immunosuppressive regimen, and receive belumosudil following the kidney transplant. Immunosuppression taper will be stopped and/or immunosuppression will be resumed for any of the following conditions:
  (1) loss of chimerism 2) clinical or pathological evidence of acute rejection and (3) clinical or pathological evidence of graft vs host disease.
  Interventions: Combination Product: Donor CD34+, CD3+. and belumosudil

INTERVENTIONS:
Combination Product: Donor CD34+, CD3+. and belumosudil — Immediately after living donor kidney transplantation, subjects will begin a conditioning regimen of rATG and total lymphoid irradiation. An infusion of at least 8 X106 donor CD34 cells/kg recipient weight and of at least 10 X106 donor CD3 cells/kg recipient weight will then be given. A triple immunosuppressive regimen of tacrolimus, corticosteroids, and mycophenolate will be utilized.
  Corticosteroids will be given on a tapering schedule from day 0 through the first four months. Tacrolimus will be given on a tapering schedule from day 1 through month 18. Mycophenolate will be given at a fixed dose from day 11 through month 12.
  Subjects will receive belumosudil 200 mg by mouth daily from day 28 following the kidney transplant through month 24.

SUMMARY:
This study seeks to determine if administration of the drug belumosudil (KD025) will be safe and improve transplant tolerance in subjects undergoing combined Human Leukocyte Antigen (HLA) single haplotype-matched related or 0-3 antigen (at A, B, C, DR) HLA mismatched unrelated living donor kidney and hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
The goal of achieving transplant tolerance (defined as prolonged graft survival in the absence of immunosuppression) has long been the aspiration of transplant physicians and researchers. Transplant tolerance may be achieved reliably and safely in HLA identical subjects undergoing combined living donor kidney and hematopoietic stem cell utilizing a conditioning regimen of Total Lymphoid Irradiation (TLI) and Rabbit anti-thymocyte globulin (rATG). However, the same treatment regimen has not been successful in allowing recipients of HLA single haplotype matched allografts to be completely withdrawn from immunosuppression in spite of increasing the dose of infused cluster of differentiation (CD) 34 and CD3 cells. This study seeks to determine the safety and efficacy of administering the investigational agent belumosudil to single haplotype- matched or HLA mismatched (0-3 antigen mismatch at HLA A, B, C, DR) subjects undergoing combined kidney and hematopoietic stem cell transplantation conditioned with TLI/rATG. Belumosudil has been shown to be highly active when used in the treatment of steroid refractory chronic graft vs host disease. We hypothesize that belumosudil (KD025) may increase mixed donor chimerism and lead to greater transplant tolerance due to its demonstrated ability to increase the numbers and function of regulatory T cells.

The summary of the treatment plan is as follows:

Immediately after living donor kidney transplantation, subjects will begin a conditioning regimen of rATG and TLI. An infusion of at least 8 X10^6 (target ≥ 10 X 10^6) donor CD34 cells/kg recipient weight and of at least 10 X10^6 (target 100 X10^6) donor CD3 cells/kg recipient weight will then be given. A triple immunosuppressive regimen of tacrolimus, corticosteroids, and mycophenolate will be utilized.

Corticosteroids will be given on a tapering schedule from day 0 through the first four months. Tacrolimus will be given on a tapering schedule from day 1 through month 18.

Mycophenolate will be given at a fixed dose from day 11 through month 12. Subjects will receive belumosudil 200 mg by mouth daily from day 28 following the kidney transplant through month 24. At serial time points, (1) chimerism will be measured in recipient whole blood and leukocyte subsets (2) graft function will be monitored (3) protocol biopsies of the graft will be obtained and (4) a T cell subsets from the peripheral blood including regulatory T cells will be measured.

Immunosuppression taper will be stopped and/or immunosuppression will be resumed for any of the following conditions:

(1) loss of chimerism (2) clinical or pathological evidence of acute rejection and (3) clinical or pathological evidence of graft vs host disease.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Age 18 and older
2. Receiving an HLA single haplotype-matched related living donor or 0-3 antigen (at A, B, C, DR) HLA mismatched unrelated living donor combined kidney and hematopoietic stem cell transplant (the first six subjects will be HLA single haplotype-matched; the final two subjects may be either HLA single-haplotype-matched or 0-3 antigen (at A, B, C, DR) HLA mismatched)
3. Agreement to participate in the study and ability to give informed consent
4. Meets institutional criteria for kidney and allogeneic hematopoietic stem cell transplant
5. Resides or is willing to stay within 3 hours distance from University of California, Los Angeles Medical Center by ground transportation for the first six months post-kidney transplant
6. No known contraindication to administration of rATG or radiation
7. If a patient is a female of reproductive potential (i.e. no documented absence of ovaries or uterus, history of tubal ligation, or post-menopausal status) patient must be confirmed not pregnancy by a serum or urine pregnancy test and must agree to practice a reliable form of contraception including hormonal treatments, barrier methods or intrauterine device for duration of the study
8. Males of reproductive age must consent to use reliable and effective methods to avoid pregnancy
9. Karnofsky Performance Score (KPS) ≥ 70
10. Adequate cardiac function defined as left ventricular ejection fracture (LVEF) ≥ 40% by Multi Gated Acquisition (MUGA) scan or echocardiogram
11. Adequate pulmonary function defined as FVC and DLCO of ≥ 50% of predicted
12. Adequate liver function defined as total bilirubin ≤ 1.5 times the upper limit of normal and AST/ALT ≤ 2.0 times the upper limit of normal
13. Adequate social support based on evaluation by the UCLA renal transplant team licensed clinical social worker
14. Negative test for COVID 19 by RT -PCR and/or have received COVID 19 vaccinations. Subjects who have not received their COVID-19 vaccination may be enrolled on the trial based on clinical judgement.

Recipient Exclusion Criteria:

1. ABO incompatibility with donor
2. Previous solid organ transplant
3. Multi-organ transplantation
4. Previous treatment with rATG or a known allergy to rabbit proteins
5. Previous treatment with belumosudil (KD025)
6. History of active malignancy within the past 5 years with the exception of:

   1. Low risk cancer on active surveillance
   2. Malignancy treated with curative intent with no known active disease >2 years before the first dose of study treatment and of low potential risk of recurrence
   3. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   4. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ, and DCIS)
7. Pregnant (confirmed by urine or serum pregnancy test) or lactating
8. Leukopenia (with a white blood cell count < 3,000/µL) or thrombocytopenia (with a platelet count < 100,000/µL)
9. INR and/or PTT ≥ 1.5X upper limits of institutional normal
10. Positive HLA DSA
11. Active bacterial, fungal, mycobacterial, or viral infection (including active hepatitis B and/or C, or West Nile Virus)
12. Seropositivity for HIV 1, HIV 2, HTLV-1 or HTLV-II
13. Renal disease with high risk of recurrence (i.e., focal segmental glomerulosclerosis)
14. Advanced hepatic fibrosis or cirrhosis
15. Congestive heart failure, symptomatic coronary artery disease, and/or uncontrolled cardiac arrhythmia
16. Active extra-renal autoimmune disease requiring immunosuppression
17. Neuropsychiatric or medical illness that precludes the ability to give informed consent and/or places the patient as high risk for non-compliance with the safety monitoring requirements of the study
18. May not have received immunosuppressive medications within one year of the study treatment. Use of corticosteroids prescribed for a time-limited indication (</= 4 weeks) and stopped at least 4 weeks before the kidney transplant is acceptable.
19. May not have received immunotherapy or immunomodulatory drugs such as immune checkpoint inhibitors, tumor necrosis factor inhibitors, rituximab, intravenous immune globulin, and interleukin-2 within one year of the study treatment
20. Current or active abuse of alcohol and/or drugs within the last 6 months
21. Body Mass Index (BMI) ≥ 40
22. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
23. ESRD patients with the following etiologies

    1. Autoimmune disease including lupus
    2. Vasculitis involving the kidney (such as Wegener's Granulomatosis
    3. Thrombotic Thrombocytopenic Purpura
    4. Alport's syndrome (due to increased risk of developing post-transplant Anti-Glomerular Basement Membrane Disease (Anti-GBM Disease))
24. HgbA1c ≥10
25. Prior history of radiation therapy
26. History of ≥ 20 pack per year smoking. a. Patients must be abstinent from tobacco use for ≥ 6 months prior to transplantation

Donor Inclusion Criteria:

1. Age 18 or older
2. HLA single haplotype-matched related living donor or 0-3 Antigen (at A, B, C, DR) HLA mismatched unrelated living donor
3. Meets institutional criteria for living kidney and allogeneic HSPC transplant donation
4. Medically fit to tolerate peripheral blood apheresis, including

   1. Weight ≥ 110 pounds
   2. Hemoglobin ≥ 11
   3. White blood cell count ≥ 3,000/µL
   4. Platelets ≥ 120,000/µL
5. Normal serum chemistry and coagulation parameter studies; or, if abnormal, the changes are not considered clinically significant
6. Negative test for COVID 19 by RT -PCR and/or have received COVID 19 vaccinations. Subjects who have not received their COVID-19 vaccination may be enrolled on the trial based on clinical judgement.

Donor Exclusion Criteria

1. ABO incompatibility with recipient
2. Medically unfit to tolerate peripheral blood apheresis (small body size, poor vascular access, not a suitable candidate for placement of a central catheter, etc.)
3. Pregnant (confirmed by urine or serum pregnancy test) or lactating
4. Seropositivity for HIV 1, HIV 2, HTLV-I or HTLV-II
5. Active bacterial, fungal, mycobacterial or viral infection (including active hepatitis B and/or C, West Nile Virus)
6. Psychiatric, addictive, neurological, or other disorder that compromises ability to give true informed consent for participation in this study
7. History of active malignancy within the past 5 years with the exception:

   1. Adequately managed malignancy within the past two years with low risk of recurrence may be acceptable as per clinician discretion
   2. Adequately managed non-melanoma skin cancer
   3. Adequately managed carcinoma in situ e.g., cervical cancer in situ, and DCIS
8. No current or recent use of oral anti-coagulants. (For the purpose of this study, recent is defined as less than 60 days prior to apheresis). Aspirin and non-steroidal anti-inflammatory drugs must be stopped 14 days prior to apheresis.
9. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Determine impact of treatment regimen on patient and kidney allograft survival | 12 months
  Measure percentage of patients alive and percentage of patients with a functioning graft at 12 months

SECONDARY OUTCOMES:
Determine probability of successful withdrawal of immunosuppression | 18 months
  Measure percentage of patients who are successfully withdrawn from mycophenolate at 12 months and from tacrolimus at 18 months
Determine risk of kidney allograft rejection | 36 months
  To determine the percentage of subjects with graft rejection within 36 months post-hematopoietic stem/progenitor cell infusion defined as (1) meets Banff criteria for rejection on biopsy performed to confirm clinical suspicion of rejection or (2) clinical suspicion of rejection demonstrating response to corticosteroids in absence of biopsy when confirmatory biopsy contraindicated or declined.
Determine risk of acute and/or chronic graft vs host disease | 36 months
  To determine percentage of patients who develop acute and/or chronic graft vs host disease within 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided